CLINICAL TRIAL: NCT05166174
Title: Lower Uterine Segment at the Next Pregnancy Following a Cesarean Section With Barbed Suture: an Observational Prospective Comparative Study
Brief Title: Lower Uterine Segment Following a Cesarean Section With Barbed Suture
Acronym: BARB-LOWSEGM
Status: Completed | Type: Observational
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, Clinical professor, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: BARB-LOWSEGM
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Cesarean Wound; Dehiscence; Cesarean Section Complications
Keywords: barbed suture; uterine lower segment; cesarean section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant women who underwent previous cesarean section with barbed suture: This group includes pregnant women, who underwent a previous cesarean section. During the previous surgical procedure, the hysterotomy was closed by using barbed suture ("Fish-bone suture").
  Interventions: Procedure: Transvaginal ultrasound in the third trimester pregnancy
- Pregnant women who underwent previous cesarean section with conventional smooth suture: This group includes pregnant women, who underwent a previous cesarean section. During the previous surgical procedure, the hysterotomy was closed conventional smooth suture.
  Interventions: Procedure: Transvaginal ultrasound in the third trimester pregnancy

INTERVENTIONS:
Procedure: Transvaginal ultrasound in the third trimester pregnancy — Ultrasonographic transvaginal exam in patients at third trimester pregnancy (34-38 weeks of gestation)

SUMMARY:
This aim of this study is to investigate the LUS in the pregnancy following a previous cesarean section with the use of barbed or conventional smooth suture.

DETAILED DESCRIPTION:
To better assess the risk of uterine rupture, some authors have proposed sonographic measurement of lower uterine segment (LUS) thickness near term, assuming that there is an inverse correlation between LUS thickness and the risk of uterine scar defect. Recently, barbed suture has been employed for closing uterine wall after cesarean section, demonstrating the reduction of closure time of the uterine incision and estimated blood loss. Until now, the impact of barbed suture in future pregnancies has not been investigated.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* being undergone a previous elective cesarean section at term of pregnancy (more than 37 weeks of gestation), in which barbed or conventional smooth suture was used for closing anterior uterine wall

Exclusion Criteria:

* having done more than one cesarean section
* having done a previous urgent cesarean section
* having done previous uterine surgical procedures with exception than one cesarean section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who underwent a previous elective cesarean section at term of pregnancy, during which the anteriore uterine wall was closed by using barbed or conventional smooth suture
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic measure of lower uterine segment thickness | 34-38 weeks following study enrollment
  Measure of lower uterine thickness (mm) at transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, Principal Investigator — Piazza della Vittoria 14, Genoa, Italy
Locations (1):
- Piazza della Vittoria 14, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jastrow N, Chaillet N, Roberge S, Morency AM, Lacasse Y, Bujold E. Sonographic lower uterine segment thickness and risk of uterine scar defect: a systematic review. J Obstet Gynaecol Can. 2010 Apr;32(4):321-327. doi: 10.1016/S1701-2163(16)34475-9. PMID 20500938
- [Background] Alessandri F, Evangelisti G, Centurioni MG, Gustavino C, Ferrero S, Barra F. Fishbone double-layer barbed suture in cesarean section: a help in preventing long-term obstetric sequelae? Arch Gynecol Obstet. 2021 Sep;304(3):573-576. doi: 10.1007/s00404-021-06121-8. PMID 34146146